CLINICAL TRIAL: NCT01384123
Title: Rehabilitation in Pulmonary Sarcoidosis: a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0019-11-MMC
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Sarcoidosis
Keywords: stable pulmonary sarcoidosis with no change in medication during the last 3 months/
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sarcoidosis is a heterogeneous multisystem disorder of unknown etiology which often presents with bilateral hilar lymphadenopathy, pulmonary infiltration and ocular and skin lesions. In addition to possible changes in forced vital capacity (FVC) and carbon monoxide transfer factor (TLCO), a higher prevalence of clinical depression, reduced health status and exercise intolerance have been observed in patients with sarcoidosis.

Reduced health status has been related to decreased pulmonary function, depressive symptoms, and to respiratory muscle weakness. Exercise capacity is believed to be limited by dyspnea, an insufficient heart rate response, decreased arterial oxygen tension during exercise, excessive and inefficient ventilation and by respiratory muscle weakness.

In the past, exercise capacity was shown to be limited by skeletal muscle weakness in patients with chronic pulmonary or cardiac disease. 67% of the sarcoidosis patients studied by Miller et al terminated their peak exercise test due to "leg complaints". Skeletal muscle weakness is therefore still assumed to be present in patients with sarcoidosis.

Treatment with oral corticosteroids, clinical symptoms of depression, myositis, self-reported complaints of fatigue and high circulating levels of tumour necrosis factor-α (TNF-α) are all present in patients with sarcoidosis and can all affect skeletal muscle force and exercise capacity. Additionally, low levels of circulating insulin-like growth factor I (IGF-I), which can be induced by high levels of TNF-α, and high circulating levels of interleukin (IL)-6 and IL-8 (CXCL8) have been associated with skeletal muscle weakness. These interleukins are part of the current concept of the immunopathogenesis of sarcoidosis16 and may be raised in patients with stable sarcoidosis.

Recent studies have shown that pulmonary rehabilitation program can lead to improve in the health status and anxiety among patients with chronic obstructive lung disease .However, no study has evaluated the role of pulmonary rehabilitation among patients with sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Stable pulmonary sarcoidosis with no change in medication during the last 3 months.

Exclusion Criteria:

* Any significant other pulmonary and\or co-morbidity that can affect exercise tolerance.
* Chronic steroid treatment more than 5 mg/day.
* Previous lung surgery.
* Advanced heart failure (NYHA III-IV )
* Malignancy during the last 3 years

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty consecutive Pulmonary sarcoidosis patients who are treated at the outpatient interstitial lung disease clinic in MEIR Medical Center.
  Pulmonary Sarcoidosis will be diagnosed according to the latest ATS/ERS/WASOG statement on sarcoidosis.1 Diagnosis of pulmonary sarcoidosis. The morphologic diagnosis of pulmonary sarcoidosis relies on three main findings: the presence of tight, well-formed granulomas and a rim of lymphocytes and fibroblasts in the outer margin of granulomas; perilymphatic interstitial distribution of granulomas (which allows transbronchial biopsies to be used as sensitive diagnostic tools); and exclusion of an alternative cause
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Improvment in 6 minute walking distance and VO2/KG max following pulmonary rehabilitation. | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel